CLINICAL TRIAL: NCT06608589
Title: CONSTELLATIONS Living Lab: Development, Implementation and Evaluation of a Patient-oriented Quality Improvement Program Targeting Care Transitions of Older Adults Living with Major Neurocognitive Disorders and Their Caregivers.
Brief Title: CONSTELLATIONS Living Lab: Improving the Care Transitions of Older Adults Living with Neurocognitive Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: CISSS de Chaudière-Appalaches (Other Government); Institut national d'excellence en santé et service sociaux (Unknown)
Responsible Party: Principal Investigator, Patrick Archambault, Patrick Archambault, MD, MSc, FRCPC. FRQS Senior Clinical Research Scholar. Professor, Department of Family Medicine and Emergency Medicine Department of Anesthesiology and Intensive Care, Université Laval., Laval University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-968, SIRUL 134632
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer Disease; Dementia; Neurocognitive Decline
Keywords: Quality improvement; Older adults; Learning Health Systems; Implementation science; Health care utilisation; Knowledge translation; Context adaptation; Care transitions; Burden of care; Emergency Department; Home care; Family medicine; Data management; Patient-oriented research; Participatory research; Living Lab; Health services; Neurocognitive disorders; Sustainability; Scale-up
MeSH Terms: conditions — Alzheimer Disease; Dementia; Emergencies; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: This study employs a mixed-methods, multilevel, quasi-experimental design with a pre-post evaluation to assess the impact of the CoMPAS+ MNCD Program intervention.
  Micro level: Quantitative and qualitative assessment of the impact of the CoMPAS+ MNCD Program on the patient reported experience in care transitions.
  Meso level (behaviour): Quantitative assessment of the intention of participating health care professionals to apply best practices in care transitions of patients living with a MNCD.
  Meso level (organisational): Quantitative and qualitative assessment of the implementation process, sustainability factors and scaling potential of the Program.
  Macro level: Comparison of administrative performance indicators between the arms and the control population (non participating LSNs in the greater Chaudière-Appalaches region and other socio-sanitary regions in the province of Quebec)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Local Services Network (LSN) Alphonse-Desjardins (Experimental): The local services network (LSN) Alphonse-Desjardins is set in a urban region with the most important community hospital of the greater region of Chaudière-Appalaches. The CoMPAS+ TNCM workshops (intervention) in the LSN Alphonse-Desjardins will be conducted with health professionals and caregiver partners from the FMG of Lévis (GMF-U de Lévis), the home support services team, and the emergency department of the Hotel-Dieu de Lévis. The population that will be recruited to evaluate the impact of the intervention will have either 1) received home care services within the last 6 months before the intervention; 2) visited the emergency department of Hotel-Dieu de Lévis within the last 6 months before the intervention; or 3) consulted with their primary health care team within the last 6 months before the intervention.
  Interventions: Other: CoMPAS+ MNCDs Program - Quality improvement program targeting the care transitions of patients living with a major neurocognitive disorder and their caregivers
- Local Services Network (LSN) Bellechasse (Experimental): The local services network (LSN) of Bellechasse is set in a rural area. The population requiring urgent medical care are lead to Hotel-Dieu de Lévis (45 km, Alphonse-Desjardins) or Hopital de Montgagny (30 km, Montmagny-L'Islet). The CoMPAS+ TNCM workshops (intervention) in the LSN of Bellechasse will be conducted with health professionals and caregiver partners from the FMG Rive de l'Etchemin (GMF Rive de l'Etchemin) which comprises the organisational merging of 2 medical clinics. Will also participate in the workshops members the home care team. The population that will be recruited to evaluate the impact of the intervention will have either 1) received home care services within the last 6 months before the intervention; 2) visited one of the 2 emergency departments (Hotel-Dieu de Lévis or Hopital de Montmagny) within the last 6 months before the intervention; or 3) consulted with their primary care team within the last 6 months before the intervention.
  Interventions: Other: CoMPAS+ MNCDs Program - Quality improvement program targeting the care transitions of patients living with a major neurocognitive disorder and their caregivers
- Local Services Network (LSN) Montmagny-L Islet (Experimental): The local services network (LSN) Montmagny-L'Islet is set in a semi-urban region with a small community hospital. The CoMPAS+ TNCM workshops (intervention) in the LSN Montmagny-L'Islet will be conducted with health professionals and careviver partners from the FMG of Montmagny (GMF de Montmagny) which comprises the organisational merging of 5 different medical clinics in the region. Will also participate in the workshops are healthcare professionals from the home care services team, and from the emergency department of the Hopital de Montmagny. The population that will be recruited to evaluate the impact of the intervention will have either 1) received home care services within the last 6 months before the intervention; 2) visited the emergency department of Hopital de Montmagny within the last 6 months before the intervention; or 3) consulted with their family doctor within the last 6 months before the intervention.
  Interventions: Other: CoMPAS+ MNCDs Program - Quality improvement program targeting the care transitions of patients living with a major neurocognitive disorder and their caregivers

INTERVENTIONS:
Other: CoMPAS+ MNCDs Program - Quality improvement program targeting the care transitions of patients living with a major neurocognitive disorder and their caregivers — COMPAS+ is a collaborative approach to improving healthcare quality. It brings together around 30 individuals, including healthcare professionals, deciders, and patient partners, to identify improvement goals, develop action plans, and enhance the prevention and management of chronic diseases. In this study, the investigators adapt COMPAS+ to focus on improving care transitions for patients with major neurocognitive disorders (MNCDs) and their caregivers. Through reflective workshops and collaborative problem-solving, this diverse group will identify best practices and create action plans to enhance care quality.

SUMMARY:
The prevalence of major neurocognitive disorders (MNCDs), particularly Alzheimer's disease, among older adults is increasing. These individuals and their caregivers often face challenges due to inefficient and poorly coordinated care transitions, negatively impacting patients, caregivers, healthcare professionals, and the healthcare system itself. To address this, the Quebec Ministry of Health and Social Services has released Phase 3 of its Ministerial Guidance on Major Neurocognitive Disorders, aiming to enhance care coordination between primary healthcare professionals and those living with MNCDs and their caregivers.

Quebec's healthcare system comprises various organizations providing care and services to individuals with MNCDs. Each organization faces unique challenges hindering improvement initiatives. However, common obstacles persist: inadequate communication systems for sharing vital information, lack of access to data for measuring care transition quality, and the absence of patient/caregiver satisfaction assessments to inform service enhancements. Additionally, organizations require support in managing change.

This need for improvement, coupled with the aspiration for a patient-centered learning health system (LHS), motivated the Institut national d'excellence en santé et services sociaux (INESSS), the Centre intégré de santé et de services sociaux de Chaudière-Appalaches (CISSS CA), and the research team to collaborate on adapting a proven continuous improvement program: the CoMPAS+ MNCD Program.

The Program will involve reflecting on best practices and identifying local challenges within participating Family Medicine Groups (FMGs) to propose and implement solutions. The CONSTELLATIONS Living Lab project has been tasked with co-developing, implementing, and evaluating the Program's impact on care transitions over two years. These findings will inform decision-makers and stakeholders about the Program's adaptability to the Chaudière-Appalaches region, guiding local and provincial decision-makers on healthcare system improvements and emphasizing the importance of supporting an LHS.

DETAILED DESCRIPTION:
1. BACKGROUND

   1.1 Context

   Patients living with major neurocognitive disorders (MNCDs) often experience inadequate care transitions, a consequence of a healthcare system struggling to adapt to their unique needs. While emergency department (ED) visits by older adults, driven by chronic illnesses, acute conditions, or social challenges, can be lifesaving, they can also lead to adverse events, unplanned readmissions (10-30%), and declines in physical, functional, and cognitive abilities. This results in distress and dissatisfaction among patients, caregivers, and healthcare workers.

   Inefficient communication and information sharing between healthcare providers further complicate the care continuum, forcing older adults and their caregivers to navigate a fragmented system they may not fully understand. To address this, the Ministerial Plan on Major Neurocognitive Disorders (The Quebec Alzheimer Plan) emphasizes interprofessional collaboration within Family Medicine Groups (FMGs) to enhance diagnosis, treatment, and follow-up for individuals with MNCDs and their caregivers. Phase 3 of this plan, launched in 2021, specifically targets improving care transitions.

   In 2018, the Institut national de santé et services sociaux (INESSS), the Centre intégré de services sociaux de Chaudière-Appalaches (CISSS CA), and a research team initiated the design of a program aimed at improving healthcare transitions for those with MNCDs. Following a pandemic-related pause, they resumed work in September 2021, adapting an existing quality improvement program for implementation within FMGs in the CISSS CA region.

   1.2. CoMPAS+ Workshop Program

   The Collective for Best Practices and the Improvement of Local Care and Services+ (CoMPAS+), led by INESSS, is a Quebec program fostering a culture of continuous improvement among integrated community service stakeholders. CoMPAS+ aims to enhance the quality of prevention and follow-up for individuals at risk of, or living with, chronic diseases. Its reflective practice workshops establish the foundation for continuous improvement projects by fostering a shared understanding of challenges related to a specific issue and promoting knowledge exchange through team reflexivity.

   Workshops commence with presentations on best practices, service utilization data, experiential knowledge from stakeholders (including patients, caregivers, and professionals), and local/regional resources relevant to the targeted disease. This shared understanding enables the identification of priority challenges and subsequent reflection on potential actions to improve quality and address these challenges.

   These workshops target key individuals within Family Medicine Groups (FMGs), Local Services Networks (LSNs), and local/regional partners. Importantly, they also include users or caregiver partners selected for their commitment and ability to contribute valuable insights. While group composition varies based on context, it generally includes:
   * Users or caregivers (mandatory participation)
   * Family physicians
   * Medical specialists relevant to the targeted chronic disease
   * Nurse practitioners specializing in primary care
   * Other professionals (social workers, respiratory therapists, nutritionists, occupational therapists, special educators, etc.)
   * Community and institutional pharmacists
   * Managers
   * Other individuals deemed relevant by the community

   1.3. Levels of assessment

   The research activities outlined in this protocol focus solely on evaluating the Program's impacts. This evaluation will be conducted at multiple levels, considering the scale of application for each activity:
   1. Micro level: Assessing the impact on users and/or caregivers.
   2. Meso level: Examining the effects on the organizations involved in the co-creation, implementation, and participation in the workshops.
   3. Macro level: Evaluating the broader impact on the population.
2. OBJECTIVES

   2.1 Primary Objective (Micro Level)

   Quantitatively evaluate the impact of the Program on care transitions for patients with MNCD and their caregivers by assessing their perceived quality of care and services from the primary care team.

   2.2 Secondary Objectives (Micro Level)

   Qualitatively assess perceptions of care transition quality to understand patient and caregiver experiences.

   Evaluate the Program's impact on the quality of life for individuals with MNCD and their caregivers.

   Assess the burden of treatment (e.g., efforts to manage health and its impact on daily life).

   Evaluate the Program's impact on caregiver burden for those caring for older adults with MNCD in the CISSS CA region.

   Assess the Program's impact on emergency department visits for individuals with MNCD in participating Local Services Networks (LSNs).

   2.3 Secondary Objective (Meso Level - Workshop Participants)

   Assess the Program's influence on workshop participants' intention to implement best practices in care transitions for individuals with MNCD and their caregivers.

   2.4 Secondary Objectives (Meso Level - Organizational)

   Identify obstacles and facilitators influencing the sustainability of the Program within the CISSS CA.

   Evaluate the potential for scaling up the Program within the CISSS CA based on the current experience.

   Recommend actions to improve the feasibility, implementation, sustainability, and scalability of the Program within the CISSS CA's FMGs.

   2.5 Secondary Objectives (Macro Level)

   Compare performance indicators and their changes over time between participating FMGs in selected LSNs and control LSNs (non-participating FMGs/LSNs).

   Assess the Program's impact on emergency department visits for people with MNCD in participating LSNs compared to non-participating LSNs (control LSNs).
3. STUDY DESIGN

   To achieve the research objectives, a mixed-methods approach will be employed. The project design involves a pre-post quasi-experimental multi-level study evaluating the impact of the CoMPAS+ MNCD Program intervention. This intervention targets clusters of professionals working within the same Local Services Network (LSN) and focuses on a specific Family Medicine Group (FMG) within that LSN.
4. STUDY POPULATIONS

   4.1 Study Population for Impact Evaluation at the User and Caregiver Level (Micro Level)

   To assess the CoMPAS+ MNCD Program's impact within each participating Local Services Network (LSN), three distinct LSNs will establish three cohorts. Each cohort will consist of dyads comprising individuals living with a Major Neurocognitive Disorder (MNCD) and their caregivers. Recognizing that individuals with MNCD may face challenges participating, caregivers may represent their dyad independently.

   Individuals with MNCD: Must reside within the socio-sanitary region served by the CISSS CA.

   Caregivers: While ideally residing within the same socio-sanitary region, caregivers from other regions may also be included.

   4.2. Study Populations at the Meso Level

   Impact of workshops on participants' intentions to apply good practices: Workshop participants

   Identification of obstacles and facilitators influencing the sustainability of the Program: Workshops participants, organizers and research team.

   Evaluation of the potential for scaling up the Program: Workshops participants, organizers and research team.

   See Eligibility section for details.
5. RECRUITMENT PROCESSES

   5.1. Micro Level Recruitment (Patients and Caregivers)

   Within each of the 3 participating LSNs, participants will be recruited from three service points: Emergency Department (ED), Home Care Team (HCT), and Family Medicine Group (FMG). The following steps will be followed at each point:

   Generate Lists: Using local administrative software, generate lists of patients who have received healthcare services within the past 6 months, applying inclusion criteria.

   Verify Eligibility: Research assistants will review each potential participant's record to confirm they meet the inclusion criteria.

   Eliminate Duplicates: Compare lists across service points to remove any duplicate entries.

   Randomize Lists: Randomize the remaining lists of potential participants.

   Contact and Consent: Research assistants will attempt to contact potential participants and their caregivers by telephone (up to five attempts) to introduce the study and assess their capacity to provide informed consent. If eligible and interested, participants will be sent a participant kit (mail or email) and recontacted after 8 days to answer any questions. Consent or refusal will be documented, and verbal e-consent forms will be securely stored in the REDCap platform.

   5.2. Meso Level Recruitment (Workshop Participants)

   All workshop participants, except the research team, INESSS stakeholders, and facilitators, will be invited to participate in the research evaluating their intent to apply best practices in care transitions.

   Email Invitation: A few days before the launch workshop, an email with a personalized REDCap link will be sent to solicit participation.

   Information and Consent: An integrated REDCap form will provide details about this research component.

   Alternative Format: Paper-based consent forms and questionnaires will be available at the first workshop for those who prefer them.

   Future Participation: Participants will be invited to express interest in future research involvement after the workshops.

   5.3. Meso Level Recruitment (Sustainability and Scale-Up)

   Key individuals involved in implementing the CoMPAS+ MNCD Program will receive email invitations to participate in research on sustainability and scale-up potential.

   Information and Consent: The form will clearly explain this research aspect and ensure voluntary participation without negative consequences for refusal.

   Participation: Participants will:

   Complete an online questionnaire twice (12-15 months apart) assessing sustainability factors and scale-up potential.

   Engage in two focus groups (before and after each workshop series) to discuss questionnaire results.

   Optionally participate in up to two individual interviews to discuss sustainability and scaling further.
6. DATA COLLECTION

   6.1 Evaluation of CoMPAS+ MNCD Program Impact on Care Transitions (Micro Level)

   Cohort Formation: Three cohorts of dyads (individuals with MNCD and their caregivers) will be recruited from three service points (ED, HCT, FMG) within each of the three participating LSNs before the CoMPAS+ MNCD workshops begin (T=0).

   Data Collection: Telephone questionnaires will be administered to consenting users and caregivers. Caregivers may answer on behalf of users with MNCD if necessary. Clinical-administrative data will also be collected from users' medical records.

   Initial Interview (T=0): The first telephone interview will cover sociodemographic characteristics, quality of life, treatment burden, care quality, information and transition experiences, and trust in the care team (for users or their caregivers). Caregivers will also be interviewed about their own sociodemographic characteristics, quality of life, involvement with their loved one, and caregiver burden.

   Follow-up Questionnaires:

   Longer questionnaires: Administered at 9 and 15 months after the initial call. Shorter questionnaires: Administered at 3 and 12 months to capture recent transition experiences and maintain contact with participants.

   Data Entry: Data collected during telephone questionnaires will be entered into the REDCap platform.

   6.2 Evaluation of Workshop Participants' Intent to Apply Best Practices

   Questionnaire Completion: Participants will complete questionnaires at multiple time points: before the launch workshop (T=0), after the launch workshop (T=1), at the end of each subsequent workshop (T=2, T=3), and 6 months after the last workshop (T=6 months).

   Workshop Introduction: During the launch workshop, 10 minutes will be allocated to explain this research component, provide the link to the online questionnaire and consent form, and offer paper-based options.

   6.3 Evaluation of Program Implementation, Sustainability, and Scale-Up Potential

   Data Collection Timeframe: Data will be collected during and after Program implementation (12-15 months post-workshops) to assess changes over time.

   Questionnaire: Key actors will complete a questionnaire twice, 12-15 months apart, assessing sustainability factors and scale-up potential.

   Focus Groups and Interviews: Focus groups will discuss aggregate questionnaire results, followed by semi-structured individual interviews to explore barriers, levers, and perspectives in more depth.

   Interview Selection: Interviewees will be selected based on diverse opinions, expertise, or preference for individual discussions.
7. MEASURING INSTRUMENTS

   7.1. Questionnaires for Impact Evaluation at the User and Caregiver Level (Micro Level)

   This study employs Patient-Reported Outcome Measures (PROMs) and Patient-Reported Experience Measures (PREMs) to assess the impact of the CoMPAS+ MNCD Program on care transitions. These instruments include both generic and specific measures to evaluate various multidimensional aspects of care transition quality, such as:

   Health and health-related quality of life (EQ-5D-5L)

   Perceived quality of care provided by the primary care team (PESQ)

   User's relationship with their care team (PESQ/FCAT)

   Treatment burden and social support (MTBQ-F)

   Caregiver burden (Zarit's Scale or Burden Inventory)

   Caregiver preparedness during transitions (FCAT)

   Participant verbatim on satisfaction with recent transitions (open questions)

   Sociodemographic data

   Service utilization data

   Clinical-administrative data from medical records

   Instrument selection was based on statistical measures (reliability and validity), popularity of use, and language availability. The research team prioritized validated French questionnaires, primarily from Canada and then France. The choice of sociodemographic, clinical-administrative, and health service utilization data was informed by the team's extensive experience in longitudinal studies, particularly with older adults.

   Further details about these instruments can be found in the 'Outcome Measures' section.

   7.2. Tool for Measuring Professional Intent Following Continuing Professional Development (CPD-reaction) (Meso Level)

   The CPD-reaction questionnaire is a validated tool based on theory (including the Theory of Planned Behavior) that evaluates the impact of training activities on healthcare professionals' behavior change. It comprises 12 items grouped into 5 dimensions:

   Behavioral intent Beliefs about abilities Social influence Beliefs about consequences Moral norm

   7.3. Measurement Tools for Assessing Sustainability and Scalability Potential (Meso Level)
   1. National Health Services Sustainability Model (NHS-SM): This empirically tested theoretical framework, accompanied by measurement tools, will be used to assess factors influencing the sustainability of the Program, guiding project leaders on priority areas for action.
   2. ISSaQ-4.0 Tool: Developed from a systematic synthesis of scientific knowledge on scaling up health innovations, this tool proposes 14 components for evaluating scaling potential, including: Health problem; Scaling up; Characteristics of innovation; Strategic, political, and environmental context of scale-up; Evidence on effectiveness; Costs and benefits; Implementation fidelity; Adaptability; Coverage; Acceptability; Adoption at scale; Scaling medium; Infrastructure; Sustainability
8. SAMPLE SIZE

   The sample size calculation was based on the following factors:

   Population: The number of individuals aged 65 and over living with an MNCD in the community (excluding those in long-term care facilities) within the CISSS CA socio-sanitary region as of March 31, 2021.

   Instrument: Validation parameters of the Physician Enabling Skills Questionnaire (PESQ).

   Study Design: Longitudinal follow-up of the same participants with questionnaires before and after the workshops and action plan implementation, necessitating a sample size calculation based on the difference of two matched averages.

   Statistical Parameters: Alpha = 0.05, power = 0.80, bilateral assumption.

   Modifiable Parameters: The clinically significant effect size of the action plan chosen by the continuous improvement team and the correlation between repeated measurements in the same individuals over time.

   Measurement Points: Three PESQ collection points at specific time points (T=0, T=9 months, T=15 months).

   Estimated Sample Size: Based on these parameters, an estimated sample size of 94 dyads per LSN would be sufficient to detect a clinically significant variation of 6.8 PESQ points.
9. DATA ANALYSIS

   1. Micro Level Analysis

      Descriptive Analyses: Basic socio-demographic data will be summarized using descriptive statistics (e.g., means, medians, frequencies, percentages).

      Bivariate Analyses: Potential associations between selected variables and primary/secondary outcomes will be explored using bivariate analyses (e.g., t-tests, chi-square tests, correlation analyses).

      Comparative Analyses: Repeated measures (pre- and post-intervention) will be compared within each LSN cohort using appropriate statistical tests (e.g., paired t-tests, Wilcoxon signed-rank tests).

      Sub-cohort Analysis: Comparative analyses will also be performed on sub-cohorts based on recruitment points (ED, HCT, FMG), adjusting for basic socio-demographic variables.
   2. Meso Level Analysis

      Linear Regression: Linear regression analysis will be conducted on DPC-Reaction constructs to identify the construct with the strongest influence on the intention to apply best practices in care transitions.

      Inferential Thematic Analysis: Focus group recordings and individual interviews will undergo inferential thematic content analysis, utilizing the NHS Sustainability Model (NHS-SM) and ISSaQ-4.0 as theoretical frameworks.
   3. Macro Level Analysis

   Indicator Comparison: Under the leadership of INESSS, performance indicators will be compared between pre-workshop years (2018-2021) and post-workshop years (2023-2025) using data provided by INESSS. This will assess changes over time and potential Program impact at the population level.
10. DATA MANAGEMENT

    Data Storage:

    Personal and Sensitive Information: Sensitive data pertaining to users and caregivers will be stored securely on the CISSS CA's server.

    Other Data: All other collected data will be entered into the REDCap database, hosted by Valeria at Laval University.

    Access Control:

    REDCap Access: Access to the REDCap database will be restricted to a limited number of research assistants and managed by the project's research coordinators.

    Full Dataset Access: Only project coordinators, the REDCap manager, and the data analysis team will have access to the complete dataset within REDCap.

    Study Staff List: A list detailing study staff members and their assigned tasks will be maintained in the project's regulatory binder, which will be stored securely under lock and key at the CISSS CA Research Centre. This list will also be submitted to the research ethics board and will be regularly updated.
11. ETHICS

    This project was approved by the Research Ethics Board of the CISSS CA, Nagano - 2023-968, SIRUL 134632
12. FUNDING

    This project was funded by the Fonds de recherche du Québec - Santé
13. CONFLICT OF INTEREST

The researcher involved in this study report having no conflict of interest.

ELIGIBILITY:
Study population for the evaluation of the impact of the CoMPAS+ MNCD Program on the care transitions of patients living with MNCD and their caregivers (Micro level)

Inclusion criteria:

* Be 65 years of age or older;
* Be living with a major neurocognitive disorder in the process of clinical evaluation or already diagnosed;
* Reside in the socio-sanitary region of the CISSS CA;
* Be able to consent independently to research (for users without caregivers at the beginning of their illness);
* Reside at home or in a retirement home or in an intermediate residence or a family-type resources;
* Consent to the research team collecting data in their medical records (FMG Electronic Medical Record (EMR) when accessible, Hospital Electronic Patient Record (EPR) when accessible, etc.).

OR

* Be the caregiver of a person 65 years of age and older living with a major neurocognitive disorder in the process of clinical evaluation or already diagnosed;
* The person being cared for must reside in the socio-sanitary region of the CISSS CA;
* Consent to the research team collecting data from the medical records of the person being cared for (FMG Electronic Medical Record (EMR) when accessible, Hospital Electronic Patient Record (EPR) when accessible, etc.);
* Be able to consent independently to research.

Exclusion criteria:

* Users living with major neurocognitive disorder under 65 years of age;
* User living in a provincial long-term care facility at the time of recruitment;
* User 65 years of age and older living with a major neurocognitive disorder, unable to consent independently to research, without a caregiver, or without a caregiver able to consent independently to research;
* Users aged 65 and over living with a major neurocognitive disorder, residing in a territory other than that of the CISSS CA;
* User refusing to consent to the collection of data in their medical records; OR
* Caregiver of a user living with a major neurocognitive disorder who does not reside in the CISSS CA territory or who is not 65 years of age or does not live at home, in a retirement home or in an IR or who died before the start of the study (T=0).
* Caregiver refusing to consent to the collection of data in the medical records of the person being cared for.

Study population for the assessment of the intention to apply best practices of CoMPAS+ MNCD workshop participants (Meso level)

Inclusion criteria:

● Be a participant in the CoMPAS+ MNCD workshops and be part of at least one of the following categories of participants:

* Health professionals working in a CISSS CA health facility or with a community organization;
* CISSS CA decision-makers or local managers;
* Community service representative (e.g., Alzheimer's Society, L'APPUI);

Exclusion criteria:

* Research team members
* Workshop facilitators
* INESSS professionals
* Users and partner caregivers
* Person unable to consent
* Person refusing to consent

Study population for the evaluation of the potential to scale-up and sustainability of the CoMPAS+ MNCD Program within the CISSS CA (Meso level)

Inclusion criteria

● Be part of one of the following categories of actors and be involved in the implementation of the CoMPAS+ MNCD Program:

* Health professionals working at the CISSS CA or in the community participating in the CoMPAS+ MNCD workshops;
* CISSS CA decision-makers;
* Users and partner caregivers;
* Community service representatives (e.g., Alzheimer's Society, L'APPUI);
* Members of the research team (except the person in charge of this component (Laetitia Bert), Alexander Cornea (research assistant), Martyne Audet (scientific coordinator), Clémence Dallaire, André Côté, Félix Pageau, Catherine Paquet);
* Research coordinator responsible for the involvement of partner users in the conduct of the workshops (Émilie Côté);
* INESSS professionals;
* Workshop facilitators
* Representative of the Ministry of Health and Social Services (MSSS).

Exclusion criteria

* Person unable to consent;
* A person refusing to consent;
* Member of the research team responsible for carrying out this part of the study or by the scientific coordination of this project (Laetitia Bert, Alexander Cornea, Martyne Audet (scientific coordinator), Clémence Dallaire, André Côté, Félix Pageau, Catherine Paquet).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Perceived quality of care: The variation in the Physician Enabling Skills Questionnaire (PESQ) scores. | Between T=0 and T=15 months with an intermediate measure at T=9 months.
  The PESQ is a 34-item scale with six subscales, used to assess the ability of family physicians to empower their patients. Total scores range from 34 to 170, with higher scores indicating greater patient autonomy facilitation. The PESQ aligns with recommendations from systematic reviews for improving care transitions, emphasizing patient and caregiver participation, provider empowerment, and decision-maker support for incremental change. This questionnaire demonstrates adequate internal consistency and has been validated in French within Quebec.
  Pre-Post Comparison: Scores will be compared to identify statistically significant changes from the patient's perspective. A variation of 6.8 PESQ points between T=0 and T=15 months will be considered significant.
  Subgroup Comparisons: Scores will be analyzed across subgroups based on recruitment points (ED, HCT, FMG) to explore any differences in perceived care quality related to the point of initial contact.

SECONDARY OUTCOMES:
Quality of life: The variation in the EQ-5D-5L questionnaire scores. | Between T=0 and T=15 months, with an intermediate measure at T=9 months.
  The EQ-5D-5L is a widely-used instrument for assessing both health status and health-related quality of life.This standardized tool evaluates five key dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Within each dimension, individuals indicate their level of severity across five response options, allowing for a nuanced understanding of their health state.
  Primary Comparison: Pre-intervention (T=0) vs. Post-intervention (T=15 months) to assess the overall impact of the CoMPAS+ MNCD Program.
  Secondary Comparisons: Changes between T=0 and T=9 months, and between T=9 months and T=15 months to track the trajectory of changes over time.
  Subgroup Analyses: Changes between different subgroups (e.g., recruitment points: ED, HCT, FMG)
Treatment burden: The variation in the Multimorbidity Treatment Burden Questionnaire-French (MTBQ-F) scores. | Between T=0 and T=15 months, with an intermediate measure at T=9 months.
  The Multimorbidity Treatment Burden Questionnaire, French-Canadian version (MTBQ-F), is a brief, 13-item tool designed to assess the treatment burden experienced by adults with chronic conditions. It identifies individuals with high treatment burdens and evaluates the impact of interventions aimed at improving their quality of care and life. MTBQ-F scores categorize treatment burden as follows: no burden (0), low (below 10), medium (10-22), and heavy (22 and over). The questionnaire boasts strong internal consistency and serves as a valuable resource for gauging the effectiveness of interventions intended to reduce treatment burden and enhance care transitions.
  Primary Comparison: Pre-intervention (T=0) scores vs. Post-intervention (T=15 months) scores to assess the overall impact of the Program on the treatment burden experienced by the older adults living with a MNCD.
  Subgroup Analyses: Changes between different subgroups (e.g., recruitment points: ED, HCT, FMG)
Caregiver burden: The variation in the Zarit questionnaire scores. | Between T=0 and T=15 months, with an intermediate measure at T=9 months.
  The Zarit Burden Interview is the most widely used standardized tool for assessing caregiver burden. It presents caregivers with a series of 12 questions (shortened version) about the challenges they face in caring for individuals with mild neurocognitive disorder (MNCD). Caregivers respond to each statement on a 5-point Likert scale, indicating their level of agreement. The total score, ranging from 0 to 48, is calculated by summing the responses to all 12 items. Higher scores reflect a heavier burden, with scores above 20 indicating a severe burden.
  Primary Comparison: Pre-intervention (T=0) scores vs. Post-intervention (T=15 months) scores to assess the overall impact of the Program on the caregivers' burden.
  Secondary Comparisons: Changes between T=0 and T=9 months, and between T=9 months and T=15 months to track the trajectory of changes over time.
  Subgroup Analyses: Changes between different subgroups (e.g., recruitment points: ED, HCT, FMG)
Qualitative content analysis of the patients and caregivers' wishes (Open-ended question). | Between T=0 and T=15 months, with an intermediate measures at T=3, 9 and 12 months.
  At the conclusion of each telephone interview, participants will be posed an open-ended question asking the participants what they would change in the healthcare system if they had a magic wand. An inductive approach will be used to iteratively develop codes and themes to categorize patient responses. This question will be asked to both patients and caregivers five times throughout their participation: at baseline (T=0), and at 3, 9, 12, and 15 months.
Variation of the intention of the workshops' participants to apply best pratices in the care for older adults living with a MNCD. | Between T=0 (pre-workshop) and 6 months post-workshops. 4 measuring points for each arm.
  The CPD-Reaction questionnaire is a validated tool grounded in theory, including the Theory of Planned Behaviour, designed to assess the impact of training activities on healthcare professionals' behavior change. It comprises 12 items organized into five dimensions: behavioral intent, beliefs about abilities, social influence, beliefs about consequences, and the moral norm. Adherence to each statement is measured on a 7-point Likert-type scale, except for social influence, which utilizes a 5-point scale.
  Primary Comparison: Pre-intervention (T=0) scores vs. Post-intervention (T=6 months)
  Secondary Comparisons: Changes between T=0 and T=6 months to track the trajectory of changes over time.
Identification of the obstacles and levers to the sustainability of the Program | T=0 and T=12 months with every arm.
  The National Health Services Sustainability Model (NHS SM) utilizes a scoring system to assess an innovation's sustainability factors. These scores then serve as the foundation for focused discussions among project leaders. In-depth, semi-structured interviews with key stakeholders subsequently delve into specific themes identified as particularly challenging during the focus groups.
  The NHS scores, while indicative of an innovation's sustainability, primarily function as catalysts for insightful discussions. These discussions, conducted in focus groups and interviews, aim to identify and comprehend the specific obstacles and levers that can be addressed to promote the long-term sustainability of the innovation.
  Primary Comparison: Qualitative comparison of obstacles and levers identified by the key stakeholders.
Program Scale-Up Potential: Variation of the ISSaQ 4.0 scores. | T=0 and T=12 months with every cohort.
  The ISSaQ-4.0 tool was developed from a systematic synthesis of scientific knowledge on the scaling up of innovative health projects. Fourteen components of scaling are proposed by this tool: 1. Health problem; 2. Scaling up; 3. Characteristics of innovation; 4. Strategic, political and environmental context of the scale-up; 5. Evidence on the effectiveness of innovation; 6. Quantifiable costs and benefits of scale-up; 7. Fidelity of the implementation of the innovation; 8. Adaptability of innovation; 9. Innovation coverage; 10. Acceptability of the innovation; 11. Adoption of innovation at scale; 12. Scaling medium; 13. Infrastructure required for scaling; 14. Sustainability.
  Primary Comparison: Pre-intervention (T=0) scores vs. Post-intervention (T=12 months)
Preparedness of caregivers to transitions: Variation of the Family Caregiver Activation in Transitions (FCAT) scores. | Between T=0 and T=15 months, with an intermediate measure at T=9 months.
  The Family Caregiver Activation in Transitions (FCAT) 10-item tool, developed by Eric A. Coleman's team, aims to foster carevivers' activation. The questionnaire underwent validation through a 3-phase approach based on a Rasch model, facilitating nuanced responses over time and for each individual item. With a person-separation reliability score of 0.84, surpassing the acceptable 0.8 benchmark for this application, the FCAT demonstrates its effectiveness in assessing and empowering caregivers during care transitions. The questionnaire has been freely translated by the research team.
  Primary Comparison: Pre-intervention (T=0) scores vs. Post-intervention (T=15 months) scores to assess the overall impact of the Program on the caregivers' preparation.
  Subgroup Analyses: Changes between different subgroups (e.g., recruitment points: ED, HCT, FMG)

OTHER OUTCOMES:
Impact of the Program at the population level: Variations of performance indicators for every LSN | Before intervention and T=18 months
  This analysis will compare performance indicators (number of ED visits, number of home care services, others) and their evolution over time between two groups:
  Participating FMGs (Family Medicine Groups) within selected Local Services Networks (LSNs).
  Control LSNs - These are LSNs with non-participating FMGs, serving as a comparison group.
  Leveraging data provided and overseen by INESSS, the impact of the CoMPAS+ TNCM workshops will be assessed by comparing performance indicators at two key time points:
  Baseline: Indicator values from the pre-workshop years (2018-2021). Post-Intervention: Indicator values in the years following the workshop (2023-2025).
  This comparison will reveal changes in performance indicators over time and any differences between the participating FMGs and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Archambault, MD, MSc, FRCPC, Principal Investigator — Laval University
Locations (1):
- Patrick Archambault, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vachon B, Desorcy B, Gaboury I, Camirand M, Rodrigue J, Quesnel L, Guimond C, Labelle M, Huynh AT, Grimshaw J. Combining administrative data feedback, reflection and action planning to engage primary care professionals in quality improvement: qualitative assessment of short term program outcomes. BMC Health Serv Res. 2015 Sep 18;15:391. doi: 10.1186/s12913-015-1056-0. PMID 26384648
- [Background] Walugembe DR, Sibbald S, Le Ber MJ, Kothari A. Sustainability of public health interventions: where are the gaps? Health Res Policy Syst. 2019 Jan 15;17(1):8. doi: 10.1186/s12961-018-0405-y. PMID 30646911
- [Background] Gugglberger L. Can health promotion also do harm? Health Promot Int. 2018 Aug 1;33(4):557-560. doi: 10.1093/heapro/day060. No abstract available. PMID 30239777
- [Background] Bergeron L, Decary S, Djade CD, Daniel SJ, Tremblay M, Rivest LP, Legare F. Factors Associated With Specialists' Intention to Adopt New Behaviors After Taking Web-Based Continuing Professional Development Courses: Cross-sectional Study. JMIR Med Educ. 2022 Jun 2;8(2):e34299. doi: 10.2196/34299. PMID 35476039
- [Background] Legare F, Borduas F, Jacques A, Laprise R, Voyer G, Boucher A, Luconi F, Rousseau M, Labrecque M, Sargeant J, Grimshaw J, Godin G. Developing a theory-based instrument to assess the impact of continuing professional development activities on clinical practice: a study protocol. Implement Sci. 2011 Mar 7;6:17. doi: 10.1186/1748-5908-6-17. PMID 21385369
- [Background] Ayivi-Vinz G, Bakwa Kanyinga F, Bergeron L, Decary S, Adisso EL, Zomahoun HTV, Daniel SJ, Tremblay M, Plourde KV, Guay-Belanger S, Legare F. Use of the CPD-REACTION Questionnaire to Evaluate Continuing Professional Development Activities for Health Professionals: Systematic Review. JMIR Med Educ. 2022 May 2;8(2):e36948. doi: 10.2196/36948. PMID 35318188
- [Background] Legare F, Borduas F, Freitas A, Jacques A, Godin G, Luconi F, Grimshaw J; CPD-KT team. Development of a simple 12-item theory-based instrument to assess the impact of continuing professional development on clinical behavioral intentions. PLoS One. 2014 Mar 18;9(3):e91013. doi: 10.1371/journal.pone.0091013. eCollection 2014. PMID 24643173
- [Background] Ajzen I. The theory of planned behaviour: reactions and reflections. Psychol Health. 2011 Sep;26(9):1113-27. doi: 10.1080/08870446.2011.613995. PMID 21929476
- [Background] Coleman EA, Ground KL, Maul A. The Family Caregiver Activation in Transitions (FCAT) Tool: A New Measure of Family Caregiver Self-Efficacy. Jt Comm J Qual Patient Saf. 2015 Nov;41(11):502-7. doi: 10.1016/s1553-7250(15)41066-9. PMID 26484682
- [Background] Hébert R, Bravo G, Girouard D. Fidélité de la traduction française de trois instruments d'évaluation des aidants naturels de malades déments. Canadian Journal on Aging / La Revue canadienne du vieillissement. 1993;12(3):324-337. doi:10.1017/S0714980800013726
- [Background] Hébert R, Bravo G, Préville M. Reliability, Validity and Reference Values of the Zarit Burden Interview for Assessing Informal Caregivers of Community-Dwelling Older Persons with Dementia. Canadian Journal on Aging / La Revue canadienne du vieillissement. 2000;19(4):494-507. doi:10.1017/S0714980800012484
- [Background] Guenette L, Turcotte V, Belanger L, Blais L, Sirois C, Lunghi C, Duncan P. Multimorbidity Treatment Burden Questionnaire (MTBQ): Translation, Cultural Adaptation, and Validation in French-Canadian. Can J Aging. 2023 Mar;42(1):126-134. doi: 10.1017/S0714980822000058. Epub 2022 May 10. PMID 35535517
- [Background] McLennan S, Kahrass H, Wieschowski S, Strech D, Langhof H. The spectrum of ethical issues in a Learning Health Care System: a systematic qualitative review. Int J Qual Health Care. 2018 Apr 1;30(3):161-168. doi: 10.1093/intqhc/mzy005. PMID 29394354
- [Background] Budrionis A, Bellika JG. The Learning Healthcare System: Where are we now? A systematic review. J Biomed Inform. 2016 Dec;64:87-92. doi: 10.1016/j.jbi.2016.09.018. Epub 2016 Sep 28. PMID 27693565
- [Background] Le Berre M, Maimon G, Sourial N, Gueriton M, Vedel I. Impact of Transitional Care Services for Chronically Ill Older Patients: A Systematic Evidence Review. J Am Geriatr Soc. 2017 Jul;65(7):1597-1608. doi: 10.1111/jgs.14828. Epub 2017 Apr 12. PMID 28403508
- [Background] Braet A, Weltens C, Sermeus W. Effectiveness of discharge interventions from hospital to home on hospital readmissions: a systematic review. JBI Database System Rev Implement Rep. 2016 Feb;14(2):106-73. doi: 10.11124/jbisrir-2016-2381. PMID 27536797
- [Background] Zhao G, Kennedy C, Mabaya G, Okrainec K, Kiran T. Patient engagement in the development of best practices for transitions from hospital to home: a scoping review. BMJ Open. 2019 Aug 5;9(8):e029693. doi: 10.1136/bmjopen-2019-029693. PMID 31383707
- [Background] Sharma AE, Knox M, Mleczko VL, Olayiwola JN. The impact of patient advisors on healthcare outcomes: a systematic review. BMC Health Serv Res. 2017 Oct 23;17(1):693. doi: 10.1186/s12913-017-2630-4. PMID 29058625
- [Background] Wilberforce, M., Challis, D., Davies, L., Kelly, M.P., Roberts, C. and Clarkson, P. (2017), Person-centredness in the community care of older people: A literature-based concept synthesis. International Journal of Social Welfare, 26: 86-98. https://doi.org/10.1111/ijsw.12221
- [Background] Rodakowski J, Rocco PB, Ortiz M, Folb B, Schulz R, Morton SC, Leathers SC, Hu L, James AE 3rd. Caregiver Integration During Discharge Planning for Older Adults to Reduce Resource Use: A Metaanalysis. J Am Geriatr Soc. 2017 Aug;65(8):1748-1755. doi: 10.1111/jgs.14873. Epub 2017 Apr 3. PMID 28369687
- [Background] Parker KJ, Hickman LD, Phillips JL, Ferguson C. Interventions to optimise transitional care coordination for older people living with dementia and concomitant multimorbidity and their caregivers: A systematic review. Contemp Nurse. 2020 Oct-Dec;56(5-6):505-533. doi: 10.1080/10376178.2020.1812416. Epub 2020 Sep 10. PMID 32820702
- [Background] Gauvin FP, McKinlay J, Markle-Reid M, Ganann R, McAiney C, Heald-Taylor G, Lavis JN. Panel summary: Engaging older adults with complex health and social needs, and their caregivers, to improve hospital-to-home transitions in Ontario. Hamilton, Canada: McMaster Health Forum, 15 November 2019.
- [Background] Hudon C, Lambert M, Almirall J. Physician Enabling Skills Questionnaire: Validation of a newly developed instrument in primary health care. Can Fam Physician. 2015 Nov;61(11):e517-23. PMID 26889507
- [Background] MEYER, John W. et ROWAN, Brian. Institutionalized organizations: Formal structure as myth and ceremony. American journal of sociology, 1977, vol. 83, no 2, p. 340-363.
- [Background] Heyland D, Cook D, Bagshaw SM, Garland A, Stelfox HT, Mehta S, Dodek P, Kutsogiannis J, Burns K, Muscedere J, Turgeon AF, Fowler R, Jiang X, Day AG; Canadian Critical Care Trials Group; Canadian Researchers at the End of Life Network. The Very Elderly Admitted to ICU: A Quality Finish? Crit Care Med. 2015 Jul;43(7):1352-60. doi: 10.1097/CCM.0000000000001024. PMID 25901550
- [Background] Haggerty JL, Reid RJ, Freeman GK, Starfield BH, Adair CE, McKendry R. Continuity of care: a multidisciplinary review. BMJ. 2003 Nov 22;327(7425):1219-21. doi: 10.1136/bmj.327.7425.1219. PMID 14630762
- [Background] van Walraven C, Taljaard M, Bell CM, Etchells E, Stiell IG, Zarnke K, Forster AJ. A prospective cohort study found that provider and information continuity was low after patient discharge from hospital. J Clin Epidemiol. 2010 Sep;63(9):1000-10. doi: 10.1016/j.jclinepi.2010.01.023. PMID 20656194
- [Background] Leppin AL, Gionfriddo MR, Kessler M, Brito JP, Mair FS, Gallacher K, Wang Z, Erwin PJ, Sylvester T, Boehmer K, Ting HH, Murad MH, Shippee ND, Montori VM. Preventing 30-day hospital readmissions: a systematic review and meta-analysis of randomized trials. JAMA Intern Med. 2014 Jul;174(7):1095-107. doi: 10.1001/jamainternmed.2014.1608. PMID 24820131
- [Background] Goncalves-Bradley DC, Lannin NA, Clemson L, Cameron ID, Shepperd S. Discharge planning from hospital. Cochrane Database Syst Rev. 2022 Feb 24;2(2):CD000313. doi: 10.1002/14651858.CD000313.pub6. PMID 35199849
- [Background] Sirois MJ, Griffith L, Perry J, Daoust R, Veillette N, Lee J, Pelletier M, Wilding L, Emond M. Measuring Frailty Can Help Emergency Departments Identify Independent Seniors at Risk of Functional Decline After Minor Injuries. J Gerontol A Biol Sci Med Sci. 2017 Jan;72(1):68-74. doi: 10.1093/gerona/glv152. Epub 2015 Sep 22. PMID 26400735
- [Background] Gill TM, Allore HG, Holford TR, Guo Z. Hospitalization, restricted activity, and the development of disability among older persons. JAMA. 2004 Nov 3;292(17):2115-24. doi: 10.1001/jama.292.17.2115. PMID 15523072
- [Background] Krumholz HM. Post-hospital syndrome--an acquired, transient condition of generalized risk. N Engl J Med. 2013 Jan 10;368(2):100-2. doi: 10.1056/NEJMp1212324. No abstract available. PMID 23301730
- [Background] Boyd CM, Landefeld CS, Counsell SR, Palmer RM, Fortinsky RH, Kresevic D, Burant C, Covinsky KE. Recovery of activities of daily living in older adults after hospitalization for acute medical illness. J Am Geriatr Soc. 2008 Dec;56(12):2171-9. doi: 10.1111/j.1532-5415.2008.02023.x. PMID 19093915
- [Background] Jencks SF, Williams MV, Coleman EA. Rehospitalizations among patients in the Medicare fee-for-service program. N Engl J Med. 2009 Apr 2;360(14):1418-28. doi: 10.1056/NEJMsa0803563. PMID 19339721
- [Background] van Walraven C, Seth R, Austin PC, Laupacis A. Effect of discharge summary availability during post-discharge visits on hospital readmission. J Gen Intern Med. 2002 Mar;17(3):186-92. doi: 10.1046/j.1525-1497.2002.10741.x. PMID 11929504
- [Background] Dudas V, Bookwalter T, Kerr KM, Pantilat SZ. The impact of follow-up telephone calls to patients after hospitalization. Dis Mon. 2002 Apr;48(4):239-48. doi: 10.1016/s0011-5029(02)90031-3. PMID 12021756
- [Background] Weaver FM, Perloff L, Waters T. Patients' and caregivers' transition from hospital to home: needs and recommendations. Home Health Care Serv Q. 1998;17(3):27-48. doi: 10.1300/j027v17n03_03. PMID 10351068
- [Background] vom Eigen KA, Walker JD, Edgman-Levitan S, Cleary PD, Delbanco TL. Carepartner experiences with hospital care. Med Care. 1999 Jan;37(1):33-8. doi: 10.1097/00005650-199901000-00006. PMID 10413390
- [Background] Harrison A, Verhoef M. Understanding coordination of care from the consumer's perspective in a regional health system. Health Serv Res. 2002 Aug;37(4):1031-54. doi: 10.1034/j.1600-0560.2002.64.x. PMID 12236382
- [Background] Grimmer KA, Moss JR, Gill TK. Discharge planning quality from the carer perspective. Qual Life Res. 2000;9(9):1005-13. doi: 10.1023/a:1016693825758. PMID 11332222
- [Background] Coleman EA, Smith JD, Frank JC, Eilertsen TB, Thiare JN, Kramer AM. Development and testing of a measure designed to assess the quality of care transitions. Int J Integr Care. 2002;2:e02. doi: 10.5334/ijic.60. Epub 2002 Jun 1. PMID 16896392
- [Background] Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003 Feb 4;138(3):161-7. doi: 10.7326/0003-4819-138-3-200302040-00007. PMID 12558354
- [Background] Dhalla IA, O'Brien T, Ko F, Laupacis A. Toward safer transitions: how can we reduce post-discharge adverse events? Healthc Q. 2012;15 Spec No:63-7. doi: 10.12927/hcq.2012.22839. No abstract available. PMID 22874449
- [Background] Qiu WQ, Dean M, Liu T, George L, Gann M, Cohen J, Bruce ML. Physical and mental health of homebound older adults: an overlooked population. J Am Geriatr Soc. 2010 Dec;58(12):2423-8. doi: 10.1111/j.1532-5415.2010.03161.x. Epub 2010 Nov 10. PMID 21070195
- [Background] Prusaczyk B, Olsen MA, Carpenter CR, Proctor E. Differences in Transitional Care Provided to Patients With and Without Dementia. J Gerontol Nurs. 2019 Aug 1;45(8):15-22. doi: 10.3928/00989134-20190530-02. Epub 2019 Jun 18. PMID 31211400
- [Background] Sakata N, Okumura Y, Fushimi K, Nakanishi M, Ogawa A. Dementia and Risk of 30-Day Readmission in Older Adults After Discharge from Acute Care Hospitals. J Am Geriatr Soc. 2018 May;66(5):871-878. doi: 10.1111/jgs.15282. Epub 2018 Feb 20. PMID 29460284
- [Background] Cadogan MP, Phillips LR, Ziminski CE. A Perfect Storm: Care Transitions for Vulnerable Older Adults Discharged Home From the Emergency Department Without a Hospital Admission. Gerontologist. 2016 Apr;56(2):326-34. doi: 10.1093/geront/gnu017. Epub 2014 Mar 28. PMID 24682396
- [Background] Smith, Brett R., and Christopher E. Stevens. 2010. "Different Types of Social Entrepreneurship: The Role of Geography and Embeddedness on the Measurement and Scaling of Social Value." Entrepreneurship &amp;amp;amp;amp;amp; Regional Development 22 (6): 575-98. doi:10.1080/08985626.2010.488405.
- [Background] Straus, S.E., Tetroe, J. and Graham, I.D. (2009). Introduction. In Knowledge Translation in Health Care (eds S.E. Straus, J. Tetroe and I.D. Graham). https://doi.org/10.1002/9781444311747.ch1
- [Background] Milat AJ, Bauman A, Redman S. Narrative review of models and success factors for scaling up public health interventions. Implement Sci. 2015 Aug 12;10:113. doi: 10.1186/s13012-015-0301-6. PMID 26264351
- [Background] Lennox L, Maher L, Reed J. Navigating the sustainability landscape: a systematic review of sustainability approaches in healthcare. Implement Sci. 2018 Feb 9;13(1):27. doi: 10.1186/s13012-017-0707-4. PMID 29426341
- [Background] Ilott I, Gerrish K, Pownall S, Eltringham S, Booth A. Exploring scale-up, spread, and sustainability: an instrumental case study tracing an innovation to enhance dysphagia care. Implement Sci. 2013 Oct 29;8:128. doi: 10.1186/1748-5908-8-128. PMID 24168667
- [Background] Levitt, Barbara, and James G. March. &amp;amp;amp;amp;#34;Organizational learning.&amp;amp;amp;amp;#34; Annual review of sociology 14.1 (1988): 319-338.
- [Background] Buchanan, D., Fitzgerald, L., Ketley, D., Gollop, R., Jones, J.L., Lamont, S.S., Neath, A. and Whitby, E. (2005), No going back: A review of the literature on sustaining organizational change. International Journal of Management Reviews, 7: 189-205. https://doi.org/10.1111/j.1468-2370.2005.00111.x
- [Background] Scheirer MA, Dearing JW. An agenda for research on the sustainability of public health programs. Am J Public Health. 2011 Nov;101(11):2059-67. doi: 10.2105/AJPH.2011.300193. Epub 2011 Sep 22. PMID 21940916
- [Background] Doyle C, Howe C, Woodcock T, Myron R, Phekoo K, McNicholas C, Saffer J, Bell D. Making change last: applying the NHS institute for innovation and improvement sustainability model to healthcare improvement. Implement Sci. 2013 Oct 26;8:127. doi: 10.1186/1748-5908-8-127. PMID 24160758
- [Background] Prince M, Bryce R, Albanese E, Wimo A, Ribeiro W, Ferri CP. The global prevalence of dementia: a systematic review and metaanalysis. Alzheimers Dement. 2013 Jan;9(1):63-75.e2. doi: 10.1016/j.jalz.2012.11.007. PMID 23305823
- [Background] Ferri CP, Prince M, Brayne C, Brodaty H, Fratiglioni L, Ganguli M, Hall K, Hasegawa K, Hendrie H, Huang Y, Jorm A, Mathers C, Menezes PR, Rimmer E, Scazufca M; Alzheimer's Disease International. Global prevalence of dementia: a Delphi consensus study. Lancet. 2005 Dec 17;366(9503):2112-7. doi: 10.1016/S0140-6736(05)67889-0. PMID 16360788
- See also: Publications du ministère de la Santé et des Services sociaux. Orientations ministérielles sur les troubles neurocognitifs majeurs - Phase 3 — https://publications.msss.gouv.qc.ca/msss/document-003346/
- See also: Publications du ministère de la Santé et des Services sociaux. Politique nationale pour les personnes proches aidantes - Reconnaître et soutenir dans le respect des volontés et des capacités d&amp;amp;amp;amp;#39;engagement. — https://publications.msss.gouv.qc.ca/msss/document-003000
- See also: Publications du ministère de la Santé et des Services sociaux. Guide de mise en oeuvre pour le déploiement des meilleures pratiques cliniques et organisationnelles dans les CISSS et les CIUSSS - Seconde phase des travaux 2016 à 2019. — https://publications.msss.gouv.qc.ca/msss/document-001825/
- See also: Projet GPS : Évaluation de l'impact de la réorganisation du travail dans les Groupes de médecine de famille (GMF) sur la Pharmacothérapie et le Soutien à l'autonomie des personnes âgées. — https://pulsar.ca/les-projets/projet/gps/fiche-complete
- See also: The National Leader In Patient and Family Centered Care Transitions Under the direction of Eric A. Coleman, MD, MPH, The Care Transitions Program provides insights and tools for how to improve quality and manage risk during care hand-overs. — https://caretransitions.org/
- See also: Implementation Practice and Science: Authors Dean Fixsen, Karen Blase, and Melissa Van Dyke summarize and synthesize advancements in implementation practice and science over the past 50 years. — https://www.activeimplementation.org/